CLINICAL TRIAL: NCT00243984
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Flexible-Dose Study to Assess the Efficacy of Topiramate for Weight Loss in Subjects With Metabolic Syndrome
Brief Title: Efficacy of Topiramate for Weight Loss in Subjects With Metabolic Syndrome
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was discontinued because of high drop out rate.
Sponsor: Northeastern Ohio Universities College of Medicine (Other)
Collaborators: Cleveland Clinic Akron General (Other); Forum Health (Industry); Aultman Health Foundation (Other); St. Elizabeth Health Center (Unknown); Mercy Medical Center (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 05005
Record Dates: First submitted 2005-10-21; First posted 2005-10-25 (Estimated); Last update posted 2007-12-10 (Estimated); Status verified 2007-12

CONDITIONS: Metabolic Syndrome X; Diabetes Mellitus, Type 2
Keywords: metabolic syndrome; type 2 diabetes; topiramate; weight loss
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus, Type 2; Weight Loss | interventions — Topiramate

INTERVENTIONS:
Drug: topiramate

SUMMARY:
The purpose of this study is to evaluate the efficacy of topiramate compared to placebo in the treatment of obesity in metabolic syndrome. Secondary objectives include topiramate and weight loss effects on lipid levels, HbA1C, insulin resistance, and blood pressure.

DETAILED DESCRIPTION:
Topiramate is an anti-convulsant which has been approved for use as adjunctive treatment for partial-onset seizures, Lennox-Gastaut syndrome, or primary generalized tonic-clonic seizures. Topiramate is currently under investigation for other disorders including binge-eating disorder.

Metabolic syndrome is a constellation of findings which includes dyslipidemia, abdominal obesity, hyperglycemia, and hypertension. Insulin resistance is believed to be the cause whereby obesity increases resistance to insulin. Weight loss in type 2 diabetics is known to reduce insulin resistance and allow for greater glycemic control. Weight loss in pre-diabetics can often forstall the development of diabetes. Additionally, aggressive blood pressure control in diabetics reduces the risk of coronary artery disease. Weight loss reduces blood pressure and is used as first line treatment for hypertension.

Comparison: Patients who meet the criteria for metabolic syndrome and prescribed topiramate will be compared with those patients who meet the same criteria and are prescribed placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Metabolic Syndrome
* BMI >/=30kg/m2
* and 3 of the 5 following criteria:

  1. Triglycerides >/=150mg/dl
  2. HDL cholesterol </=40mg/dl (men) or </=50mg/dl (women)
  3. Blood pressure > 130/85
  4. Waist circumference >/=40inches (men) or >/=35inches (women)
  5. Fasting blood glucose >/=110mg/dl or diagnosis of type 2 diabetes mellitus
* Able to give informed consent
* Diabetes Mellitus must be well controlled for the past 3 months and HbA1c </=9.0
* Hypertension must be well controlled for the past 3 months and BP <140/90
* Willing and able to take oral medication
* Female subjects must be post menopausal for 1 year, surgically sterile, or practicing an effective method of birth control; and have a negative monthly pregnancy test at screening and throughout the study.

Exclusion Criteria:

* Any person unable to take topiramate
* Renal insufficiency
* Taking medication with known serious interactions with topiramate
* History of psychosis, epilepsy or any other disease in which taking topiramate may interfere with treatment of that disease
* Positive urine drug screen
* Previous treatment with topiramate and subsequent adverse event; or concurrent treatment with topiramate
* History of nephrolithiasis
* Pregnancy or lactating
* Subjects who are members of the same household
* Currently on an exercise or diet plan
* Bariatric surgery within the past 5 years
* Clinically significant medical conditions including (but not limited to) symptomatic coronary artery disease or peripheral vascular disease, or taking nitrates; malignancy or history of malignancy within the past 5 years (except basal cell carcinoma); Impaired renal function as defined by an estimated creatinine clearance </=60ml/min; Gastrointestinal system diseases including active liver disease; ALT or AST>2 times the upper limit of normal; Pulmonary disorders; Endocrine disorders except for well controlled diabetes mellitus and hypothyroidism; Any disease or condition that compromises the function of those body systems that could result in altered absorption, excess accumulation, or impaired metabolism or excretion of topiramate.
* Subjects who in the opinion of the investigator should not be enrolled in the study because of the precautions, warnings, or contraindications sections of the topiramate package insert
* Family members of employees or investigators and employees of the investigator or study center may participate but may not serve any staff role for themselves.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2005-03; Study Completion 2007-11 (Estimated)

PRIMARY OUTCOMES:
Change in weight on days 28, 56, 84, 112, 140, 168, and 175.
Waist circumference on days 1, 84 and 168.
BMI on days 1, 84, 168, and 175.

SECONDARY OUTCOMES:
Blood pressure on days 1, 28, 56, 84, 112, 140, 168, and 175.
Complete metabolic profile on days 84 and 168.
HbA1C on days 1, 84, and 168.
Lipid profile on days 84 and 168.
C reactive protein on days 1, 84, and 168.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Whittier, MD, Principal Investigator — Northeastern Ohio Universities College of Medicine
Locations (5):
- United States (5):
  - Akron General Medical Center, Akron, Ohio
  - Mercy Medical Center, Canton, Ohio
  - Aultman Hospital, Canton, Ohio
  - Forum Health/Northside Medical Center, Youngstown, Ohio
  - St. Elizabeth Health Center, Youngstown, Ohio